CLINICAL TRIAL: NCT06418919
Title: A Prospective Evaluation of Radiofrequency Ablation in the Treatment of Relapsed Graves' Disease.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lang Hung Hin, Brian, Clinical Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 22-504
Record Dates: First submitted 2024-05-10; First posted 2024-05-17 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Relapsed Graves' Disease; Thyroid; Functional Disturbance; Radiofrequency Ablation Treatment
MeSH Terms: conditions — Graves Disease; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFA treatment (Experimental)
  Interventions: Procedure: Radiofrequency ablation treatment

INTERVENTIONS:
Procedure: Radiofrequency ablation treatment — RFA is used to ablate the entire thyroid gland

SUMMARY:
There have been previous reports of using High-intensity focused ultrasound (HIFU) as a feasible thermal ablative treatment for relapsed Graves' disease. In recent years, radiofrequency ablation (RFA) has become another promising alternative for thermal ablation of benign thyroid nodules. RFA has the advantage of avoiding a surgical scar, organ preservation and being an ambulatory procedure. It utilizes a small caliber radiofrequency electrode, which is inserted into the thyroid gland percutaneously. The active tip of the RF electrode would induce frictional heat in the surrounding tissue, causing a thermal ablative effect. The direct application of energy of RFA to tissue is different from that in HIFU, in which energy is transmitted through the skin of the participants from the transducer.

Studies of follow-up after RFA of Graves' disease have not been published. Given the previous successful experience with HIFU, the investigators would like to explore the feasibility, safety and efficacy of RFA as an alternative thermal ablation option for relapsed Graves' disease. Thus, the purpose of this prospective study is to assess the efficacy and safety of US-guided RFA for the treatment of relapsed Graves' disease.

ELIGIBILITY:
Inclusion Criteria:

* (a) age older than 18 years,
* (b) relapsed Graves' disease despite an adequate ATD treatment for 18 months or more and
* (c) absence of vocal cord immobility.

Exclusion Criteria:

* (a) patients who prefer or indicated for surgery,
* (b) head and/or neck disease preventing hyperextension of the neck,
* (c) history of thyroid cancer or other malignant tumors in the neck region,
* (d) history of neck irradiation,
* (e) moderate to severe Graves' ophthalmopatty,
* (f) large compressive goiter
* (g) pregnancy or lactation, and
* (h) any contraindication related to intravenous moderate sedation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Short term disease remission rate after a single course of RFA | 12 months
  Graves' disease remission rate after a single course of RFA
Mid term remission rate after a single course of RFA | 24 months and 36 months
  Graves' disease remission after a single course of RFA
Complication rates | 1 month
  To measure the complication rates after RFA
Change in Quality of life | 24 months, 36 months
  To examine the change in qualitfy of life with SF-12 scores in post-treatment from baseline to 24 months and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Matrix, Man Him Fung, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Cooper DS. Antithyroid drugs. N Engl J Med. 2005 Mar 3;352(9):905-17. doi: 10.1056/NEJMra042972. No abstract available. PMID 15745981
- [Background] Watanabe N, Narimatsu H, Noh JY, Yamaguchi T, Kobayashi K, Kami M, Kunii Y, Mukasa K, Ito K, Ito K. Antithyroid drug-induced hematopoietic damage: a retrospective cohort study of agranulocytosis and pancytopenia involving 50,385 patients with Graves' disease. J Clin Endocrinol Metab. 2012 Jan;97(1):E49-53. doi: 10.1210/jc.2011-2221. Epub 2011 Nov 2. PMID 22049174
- [Background] Yip J, Lang BH, Lo CY. Changing trend in surgical indication and management for Graves' disease. Am J Surg. 2012 Feb;203(2):162-7. doi: 10.1016/j.amjsurg.2011.01.029. Epub 2011 Jun 17. PMID 21683939
- [Background] Lang BH, Woo YC, Chiu KW. Two-year outcomes of single-session high-intensity focused ultrasound (HIFU) treatment in persistent or relapsed Graves' disease. Eur Radiol. 2019 Dec;29(12):6690-6698. doi: 10.1007/s00330-019-06303-8. Epub 2019 Jun 17. PMID 31209622
- [Background] Lang BH, Woo YC, Wong IY, Chiu KW. Single-Session High-Intensity Focused Ultrasound Treatment for Persistent or Relapsed Graves Disease: Preliminary Experience in a Prospective Study. Radiology. 2017 Dec;285(3):1011-1022. doi: 10.1148/radiol.2017162776. Epub 2017 Jul 20. PMID 28727542
- [Background] Kim JH, Baek JH, Lim HK, Ahn HS, Baek SM, Choi YJ, Choi YJ, Chung SR, Ha EJ, Hahn SY, Jung SL, Kim DS, Kim SJ, Kim YK, Lee CY, Lee JH, Lee KH, Lee YH, Park JS, Park H, Shin JH, Suh CH, Sung JY, Sim JS, Youn I, Choi M, Na DG; Guideline Committee for the Korean Society of Thyroid Radiology (KSThR) and Korean Society of Radiology. 2017 Thyroid Radiofrequency Ablation Guideline: Korean Society of Thyroid Radiology. Korean J Radiol. 2018 Jul-Aug;19(4):632-655. doi: 10.3348/kjr.2018.19.4.632. Epub 2018 Jun 14. PMID 29962870
- [Background] Kuo JH, Lee JA. The Adoption of Ultrasound-guided Radiofrequency Ablation of Thyroid Nodules in the United States. Ann Surg. 2021 Jan 1;273(1):e10-e12. doi: 10.1097/SLA.0000000000003930. No abstract available. PMID 33064390
- [Background] Papini E, Pacella CM, Solbiati LA, Achille G, Barbaro D, Bernardi S, Cantisani V, Cesareo R, Chiti A, Cozzaglio L, Crescenzi A, De Cobelli F, Deandrea M, Fugazzola L, Gambelunghe G, Garberoglio R, Giugliano G, Luzi L, Negro R, Persani L, Raggiunti B, Sardanelli F, Seregni E, Sollini M, Spiezia S, Stacul F, Van Doorne D, Sconfienza LM, Mauri G. Minimally-invasive treatments for benign thyroid nodules: a Delphi-based consensus statement from the Italian minimally-invasive treatments of the thyroid (MITT) group. Int J Hyperthermia. 2019;36(1):376-382. doi: 10.1080/02656736.2019.1575482. Epub 2019 Mar 26. PMID 30909759
- [Derived] Fung MHM, Luk Y, Yuen KKW, Lang BHH. The Two-Year Results of Using Radiofrequency Ablation as a Novel Treatment for Persistent or Relapsed Graves' Disease: A Prospective Study. Thyroid. 2024 Aug;34(8):1017-1026. doi: 10.1089/thy.2024.0177. Epub 2024 Jul 3. PMID 38836419
- See also: Ultrasound-guided percutaneous radiofrequency ablation for benign thyroid nodules — http://www.nice.org.uk/guidance/ipg562